CLINICAL TRIAL: NCT06656026
Title: A Open-label Phase 2 Study of ZSP1273 in Otherwise Healthy Children 2-17 Years Old With Influenza A
Brief Title: Pharmacokinetics，Safety and Efficacy of ZSP1273 in Children 2-17 Years Old With Influenza A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ZSP1273-23-17
Record Dates: First submitted 2024-10-14; First posted 2024-10-24 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-10

CONDITIONS: Influenza a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZSP1273(Arm a) (Experimental): * ≥2 ，<6 year old，dose 1 QD；5day
  * ≥6 ，<12 year old，dose 2 QD；5day
  * ≥12，≤17 year old，dose 3 QD；5day
  Interventions: Drug: ZSP1273 granules
- ZSP1273(Arm b) (Experimental): * ≥2 ，<6 year old，dose 4 QD；5day
  * ≥6 ，<12 year old，dose 5 QD；5day
  * ≥12，≤17 year old，dose 6 QD；5day
  Interventions: Drug: ZSP1273 granules

INTERVENTIONS:
Drug: ZSP1273 granules — Oral

SUMMARY:
This trial is conducted in China. The aim of the trial is to investigate safety,pharmacokinetics and pharmacodynamics of ZSP1273 granules

ELIGIBILITY:
Inclusion Criteria:

1. Subjects and their guardians who are able to understand the study and comply with all study procedures, and willing to provide written informed consent/assent prior to the predose examinations appropriately.
2. Male or female subjects aged ≥ 2 to ≤17 years at the time of signing the informed consent form.
3. Subjects with a diagnosis of influenza virus infection confirmed by all of the following:

   * Positive rapid antigen test (RAT) for influenza with nasal or throat swabs;
   * The time interval between the onset of symptoms and enrollment is 72 hours or less;
   * Fever ≥ 38ºC (axillary temperature); and at least one following respiratory symptoms associated with influenza virus infection is present

Exclusion Criteria:

1. Subjects with severe influenza virus infection；
2. Subjects with any medical history in gastrointestinal that interferes with the absorption of drugs；
3. Immunodeficiency,including malignant tumor,organ or marrow transplant,human immunodeficiency virus [HIV] infection,or patients receiving immunosuppressant therapy 3 months prior to enrollment；
4. Have received any other investigational products within 3 months prior to dosing；
5. Positive urine pregnancy test；
6. Subjects with concurrent infections requiring antimicrobial therapy；
7. Subjects who are considered inappropriate for the study by the investigator.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of ZSP1273 | DAY1~5

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | DAY1~29
Time to alleviation of influenza symptoms (duration of influenza) | DAY1~29
Percentage of subjects with virus titer detected | DAY1~29

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong, China